CLINICAL TRIAL: NCT03689491
Title: Investigating the Effects of Combining rTMS With Visual Feedback Training to Improve Movements in the Paretic Lower Limb and Gait Performance
Brief Title: The Combining rTMS With Visual Feedback Training for Patients With Stroke
Acronym: rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105TMU-TMUH-14
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2018-09

CONDITIONS: Stroke
Keywords: rTMS; visual feedback; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Outcomes Assessor
Masking Description: Single Blind (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS+visual feedback (Experimental): 10-minute rTMS and then a 30-minute visual feedback training ,3 times a week, for 4 weeks
  Interventions: Behavioral: rTMS; Behavioral: visual feedback training
- sham rTMS+visual feedback (Active Comparator): 10-minute sham rTMS and then a 30-minute visual feedback training ,3 times a week, for 4 weeks
  Interventions: Behavioral: rTMS; Behavioral: visual feedback training
- sham rTMS+traditional training (Active Comparator): 10-minute sham rTMS and then a 30-minute traditional rehabilitation training,3 times a week, for 4 weeks
  Interventions: Behavioral: rTMS; Behavioral: traditional rehabilitation

INTERVENTIONS:
Behavioral: rTMS — The EMG measured the MEPs of the anterior tibialis in response to the TMS delivered using a Magstim Rapid2 stimulator (Magstim Co, Ltd, Carmarthenshire, Wales, UK) with a 70-mm figure-8 coil (maximum power, 2.2 T) over the contralateral M1. The intensity was initially set at 100% of the machine output (MO) to determine the optimal stimulation site (hotspot). The hotspot was marked on the scalp with oil ink and recorded as x, y, in centimeters from the vertex (cz). The participants received real rTMS or sham rTMS, respectively (1 Hz, 10 min), which was before a 30-minute visual feedback training and/or traditional rehabilitation training.
Behavioral: visual feedback training — Game-based visual feedback training system and software.The system was designed to enable the subjects to perform ankle movements in multiple axes.
  Arms: rTMS+visual feedback; sham rTMS+visual feedback
Behavioral: traditional rehabilitation — 30 min traditional rehabilitation. The traditional rehabilitation programs included balance training, postural training, muscle strengthening, ambulation training and etc..
  Arms: sham rTMS+traditional training

SUMMARY:
After stroke, patients often experience motor deficits that interrupt normal lower extremity movement and gait function. Recent developments in neuroimaging have focus on the reasons why some patients recover well while some do poorly. However, there is still no consensus on the exact mechanisms involved in regaining the functions after rehabilitation. Application of repetitive transcranial magnetic stimulation (rTMS) to facilitate neural plasticity during stroke treatment has recently gained considerable attention. The possible mechanism through which rTMS acts is based on the interhemispheric competition (IHC) model, which explains that patients with stroke experience alterations in cortical excitability and exhibit abnormally high interhemispheric inhibition from the unaffected hemisphere to the affected hemisphere. The visual feedback training can improve postural control and enhance motor performance. Several rTMS studies have evaluated the lower extremity dysfunction following stroke, but few studies have explored the efficacy of applying rTMS on the lower extremities. We expect the study can help us to further exploration of the change of clinical function and cortical excitability following rTMS and visual feedback training in subjects with stroke. In addition, the results of this project will be provided for further rehabilitation programs in people with stroke.

DETAILED DESCRIPTION:
Objective: To investigate the effects of combining rTMS with visual feedback training to improve movements in the paretic lower limb and gait performance.

Methods: Thirty patients with monohemispheric after ischemic stroke will recruited and randomized into 3 groups. The group 1 received a 10-minute rTMS intervention then a 30-minute visual feedback training. The group 2 received a 10-minute sham rTMS intervention then a 30-minute visual feedback training. The group 3 received a 10-minute sham rTMS intervention then a 30-minute traditional rehabilitation training. All subjects received treatments 3 times a week for 4 weeks. The performance was assessed by a blinded assessor for two times (baseline and after 4 weeks). The outcome measures included Motor evoked potential (MEP), Fugl-Meyer Assessment-Lower Limb section(FMA-LE),Motor Assessment Score(MAS), Berg Balance Test (BBS),Time Up and Go (TUG), and Modified Barthel Index for ADL ability. Collected data will be analyzed with ANOVA test by SPSS version 20.0, and alpha level was set at 0.05. The hypothesis is combining rTMS with visual feedback training has positive effects on lower limb and gait performance among patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Monohemispheric ischemic or hemorrhage stroke
2. Subjects with first-ever stroke 3.6 months after stroke onset

4.The Brunnstrom stage of lower limb >Ⅲ 5.>23 in the mini-mental state exam 6.The Modified Ashworth Scale of lower limb <3 7.Clear consciousness can meet the relevant assessments

Exclusion Criteria:

1. Recurrent stoke
2. Severe spasticity of lower limb and difficult to perform isolative movement.
3. History of seizures or epileptic
4. Have implanted ferromagnetic devices or other magnetic-sensitive metal implants
5. Concomitant vestibular and cerebellum diseases
6. Joint contracture of lower limb/foot and other orthopedic problems
7. Subjects with severe cognitive impairment
8. Subjects with depression and/or mood disorder
9. Presence of any comorbid neurological diseases or psychological diseases

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Change of Motor evoked potential | Change from baseline to 4 weeks
  Measurement of motor evoked potential of anterior tibialis

SECONDARY OUTCOMES:
Chang of Motor Assessment Score | Change from baseline to 4 weeks
  Lower Limb motor function
Chang of Berg Balance Test | Change from baseline to 4 weeks
  standing balance
Chang of Fugl-Meyer Assessment-Lower Limb section | Change from baseline to 4 weeks
  Lower Limb section
Chang of Modified barthel index | Change from baseline to 4 weeks
  Activity of daily live ability
Chang of Time Up and Go | Change from baseline to 4 weeks
  functional ambulation

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Hsien-Lin, Master, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No